CLINICAL TRIAL: NCT05329402
Title: Clinical Trial on Performance and Safety of Disposable Powered Articulating Linear Cutter Stapler and Reloads in Total-Thoracoscopic Anatomic Lobectomy (Segmentectomy)
Brief Title: Disposable Powered Articulating Linear Cutter Stapler in Total-Thoracoscopic Anatomic Lobectomy (Segmentectomy)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fengh Medical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20256031708-BC1
Record Dates: First submitted 2022-03-31; First posted 2022-04-15 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2023-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Disposable Powered Articulating Endoscopic Linear Cutter Stapler (Experimental): Disposable Powered Articulating Endoscopic Linear Cutter Stapler
  Interventions: Device: Disposable Powered Articulating Endoscopic Linear Cutter Stapler
- ECHELON Flex Powered Articulating Endoscopic Linear Cutters (Active Comparator): ECHELON Flex Powered Articulating Endoscopic Linear Cutters
  Interventions: Device: ECHELON Flex Powered Articulating Endoscopic Linear Cutters

INTERVENTIONS:
Device: Disposable Powered Articulating Endoscopic Linear Cutter Stapler — Using the Disposable Powered Articulating Endoscopic Linear Cutter Stapler according to routine treatment
  Arms: Disposable Powered Articulating Endoscopic Linear Cutter Stapler
Device: ECHELON Flex Powered Articulating Endoscopic Linear Cutters — Using the ECHELON Flex Powered Articulating Endoscopic Linear Cutters according to routine treatment
  Arms: ECHELON Flex Powered Articulating Endoscopic Linear Cutters

SUMMARY:
To evaluate whether the anastomosis success rate of the main effectiveness evaluation indexes is not inferior to the similar products produced by Johnson & Johnson when the Fengh Disposable Powered Articulating Endoscopic Linear Cutter Stapler Used for Thoracoscopic Anatomic Lobectomy (segmentectomy)

DETAILED DESCRIPTION:
By comparing the effectiveness and safety of the disposable electric-endoscopic linear cutter stapler and cartridge (the subject product) produced by Jiangsu Fengh Medical Co., Ltd. and the similar product (electric-endoscopic linear cutter stapler with articulating head) produced by Johnson & Johnson in total-thoracoscopic anatomic lobectomy (segmentectomy), to prove that the subject product can be used for pulmonary tissue resection and anastomosis, and that the clinical trial meets the requirements of Good Clinical Practice for Medical Devices, Guidelines for Clinical Trial Design of Medical Devices and Guidelines for Technical Review of Endoscopic Stapler Registration, which can be used for product registration application.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18-70 (inclusive), with no gender limitation;
2. The subject plans to undergo thoracoscopic anatomic pulmonary lobectomy (pulmonary segment);
3. Subjects or their guardians can understand the purpose of the study, show sufficient compliance with the study protocol, and sign the informed consent.

Exclusion Criteria:

1. Subjects have contraindications of video-assisted thoracoscopy;
2. The preoperative imaging results of the subjects indicated the presence of severe pleural adhesion and significant calcified hilar lymph nodes;
3. Subjects' platelet (PLT) <60x 10%/L or INR > 1.5;
4. Subjects forced expiratory volume in 1 second (FEV1)/expected value ≤50%, or forced expiratory volume in 1 second (FEV1)/use Vital capacity (FVC)≤60%;
5. Cardiac ejection fraction ≤50%;
6. Major organ failure or other serious diseases (including clinically relevant cardiovascular diseases or within 12 months prior to enrollment) Myocardial infarction; A history of severe neurological or psychiatric illness; The presence of a serious infection before surgery that must be controlled with medication; Dissemination of activity Sexual intravascular coagulation; At high risk of blood clots);
7. The subject is a pregnant or lactating woman;
8. The subject participated in clinical trials of other drugs or devices within 1 month prior to the trial;
9. Other conditions that the researcher judged inappropriate for inclusion. .

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2020-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yusheng Shu, Principal Investigator — Northern Jiangsu People's Hospital
Locations (1):
- Disposable Powered Articulating Endoscopic Linear Cutter Stapler, Jiangyin, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Only the results of CT, routine blood test, coagulation function, fasting blood glucose, occult blood test of stool, cardiac ultrasound, lung function and digestive tract angiography were available to the participants, and other results were not shared

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 30 days
Groups:
- Disposable Powered Articulating Endoscopic Linear Cutter Stapler: The Disposable Powered Articulating Endoscopic Linear Cutter Stapler is intended for transection, resection, and/or creation of anastomoses. The instrument has application in multiple open or minimally invasive general, gynecologic, urologic, thoracic, and pediatric surgical procedures. It can be used with staple line or tissue buttressing materials. The instrument may also be used for transection and resection of liver parenchyma (hepatic vasculature and biliary structures), pancreas, kidney and spleen.
- ECHELON Flex Powered Articulating Endoscopic Linear Cutters: ECHELON Flex Powered Articulating Endoscopic Linear Cutters has application in multiple open or minimally invasive general, gynecologic, urologic, thoracic, and pediatric surgical procedures.
Period: Overall Study
Arm/Group | Disposable Powered Articulating Endoscopic Linear Cutter Stapler | ECHELON Flex Powered Articulating Endoscopic Linear Cutters
Started | 80 | 84
Completed | 79 | 83
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Disposable Powered Articulating Endoscopic Linear Cutter Stapler: The Disposable Powered Articulating Endoscopic Linear Cutter Stapler is intended for transection, resection, and/or creation of anastomoses. The instrument has application in multiple open or minimally invasive general, gynecologic, urologic, thoracic, and pediatric surgical procedures. It can be used with staple line or tissue buttressing materials. The instrument may also be used for transection and resection of liver parenchyma (hepatic vasculature and biliary structures), pancreas, kidney and spleen.
  Lung cancer surgery: Only the brand of electric cutting stapler used by different groups was different, and the rest were treated according to routine treatment
- ECHELON Flex Powered Articulating Endoscopic Linear Cutters: ECHELON Flex Powered Articulating Endoscopic Linear Cutters has application in multiple open or minimally invasive general, gynecologic, urologic, thoracic, and pediatric surgical procedures.
  Lung cancer surgery: Only the brand of electric cutting stapler used by different groups was different, and the rest were treated according to routine treatment
- Total: Total of all reporting groups
Arm/Group | Disposable Powered Articulating Endoscopic Linear Cutter Stapler | ECHELON Flex Powered Articulating Endoscopic Linear Cutters | Total
Number analyzed (Participants) | 79 | 83 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.95 (9.77) | 55.33 (8.94) | 55.14 (9.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 51 | 91
  Male | 39 | 32 | 71
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 79 | 83 | 162
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.88 (3.34) | 24.06 (3.24) | 23.97 (3.28)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Anastomosis Success
Description: The transection and anastomosis of lung tissues are performed during the operation. The device is withdrawn after successful triggering. The cutting staple line is carefully checked for integrity, air leakage and bleeding. If all staple lines are complete, without air leakage or bleeding, it is judged that the cutting and anastomosis of the device is successful. If there is persistent air leakage and bleeding at the anastomosis site, and conversion to thoracotomy is required, it is judged as device cutting and anastomosis failure.
Time Frame: During surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Disposable Powered Articulating Endoscopic Linear Cutter Stapler | ECHELON Flex Powered Articulating Endoscopic Linear Cutters
Number analyzed (Participants) | 79 | 83
Participants | 79 | 83
Statistical Analysis 1: Comparison: Disposable Powered Articulating Endoscopic Linear Cutter Stapler vs ECHELON Flex Powered Articulating Endoscopic Linear Cutters; Test type: Non-Inferiority — The non-inferiority hypothesis is tenable if the lower limit of 95% confidence interval of the difference in the primary effectiveness evaluation indicator "device cutting and anastomosis success rate" between the test group and the control group is greater than the non-inferiority critical value (-10%); p = 0.9727, Wald; Mean Difference (Final Values) = 0, 95% CI 2-sided [-0.0285 to 0.0273]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Disposable Powered Articulating Endoscopic Linear Cutter Stapler | ECHELON Flex Powered Articulating Endoscopic Linear Cutters
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/83
Serious Adverse Events (participants affected / at risk) | 10/79 | 8/83
Other Adverse Events (participants affected / at risk) | 44/79 | 54/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Disposable Powered Articulating Endoscopic Linear Cutter Stapler (N=79) | ECHELON Flex Powered Articulating Endoscopic Linear Cutters (N=83)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Right pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary artery bleeding (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aerodermectasia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thoracic wall lung hernia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Lung leak gas (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
left chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Acute cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Left lower lung with residual pulmonary atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Chylopleura (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abnormal liver function (Hepatobiliary disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Disposable Powered Articulating Endoscopic Linear Cutter Stapler (N=79) | ECHELON Flex Powered Articulating Endoscopic Linear Cutters (N=83)
constipation (Gastrointestinal disorders) | 11 (11) | 10 (10)
emesis (Gastrointestinal disorders) | 7 (7) | 7 (7)
aypnia (Nervous system disorders) | 8 (8) | 5 (6)
others (General disorders) | 18 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/02/NCT05329402/Prot_SAP_000.pdf